CLINICAL TRIAL: NCT04711018
Title: Comparison of Various Measures for Anticipating Difficult Laryngoscopy in Turkish Population: An Observational Study
Brief Title: Comparison of Various Measures for Anticipating Difficult Laryngoscopy
Acronym: COMPAD-T
Status: Completed | Type: Observational
Sponsor: Yedikule Training and Research Hospital (Other)
Collaborators: Avcılar Murat Koluk State Hospital (Unknown)
Responsible Party: Principal Investigator, Derya Ozden Omaygenc, M.D., Haseki Training and Research Hospital
Other Study IDs: HasekiTRERH
Record Dates: First submitted 2021-01-09; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Difficult Laryngoscopy
Keywords: Cephalometry; Endotracheal intubation; Ethnicity; Laryngoscopy
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group DL (+): Grade III or IV laryngeal view according to Cormack-Lehane classification
  Interventions: Diagnostic Test: Laryngoscopy
- Group DL (-): Grade I or II laryngeal view according to Cormack-Lehane classification
  Interventions: Diagnostic Test: Laryngoscopy

INTERVENTIONS:
Diagnostic Test: Laryngoscopy — The laryngoscopy is performed with the help of an appropriate size Macintosh blade. The patient's head is held in the sniffing position. External manipulation is not used for improving the view in this investigation.

SUMMARY:
Demographic features and eight diagnostic variables were evaluated for difficult laryngoscopy (DL) predictivity. These were retrognathia, presence of buck teeth, modified Mallampati test (MMT), upper lip bite test (ULBT), sternomental distance (SMD), interincisor distance (IID), thyromental distance, and neck circumference. DL was identified by Grade III-IV view during laryngoscopy according to the Cormack-Lehane (CL) classification.

DETAILED DESCRIPTION:
Creating a regression model among selected bedside tests for predicting difficult laryngoscopy )defined as Grade III or IV view during laryngoscopy according to Cormack-Lehane classification) is the primary objective. Recruiting of 145 ASA I-II adult patients who would have an elective surgery under general anesthesia were planned.

Criteria for exclusion were: a history of craniofacial surgery or restriction of cervical mobility, edentulous patients, pregnant women, patients who did not have a proper mouth opening (< 3 cm), and those who might require awake intubation or rapid sequence induction, cancellation of the surgery or change in the anesthetic strategy.

The selected tests and clinical situations were:

The presence of retrognathia (reduced temporomandibular joint-incisor distance) Buck teeth Modified Mallampati test (MMT) in the sitting position without phonation. A scale ranging between 1 and 4 points is used and scores of 3 or 4 are considered as predictors of DL. Upper lip bite test (ULBT) performed in a neutral position. ULBT is graded as 1-3 according to the extension ability of lower incisors.

Sternomental distance - The distance between the mentum and upper border of the manubrium sterni when the head is fully extended and the mouth is closed.

Thyromental distance (TMD) - The distance between mentum and the thyroid notch when the head is fully extended.

Interincisor distance (IID) - The distance between upper and lower incisors when the mouth is fully opened.

Neck circumference (NC) - It was measured at the level of the cricoid cartilage, perpendicular to the cervical axis.

The patients are premedicated with 0.03 mg/kg and oxygenated with the help of a bag-mask. Anesthesia is induced by consequent administration of 2 mcg/kg fentanyl, 1 mg/kg lidocaine, 2 mg/kg propofol, and 0.7 mg/kg rocuronium bromide thereafter. Two minutes after induction, the laryngoscopy is performed

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Candidate for elective surgery under general anesthesia

Exclusion Criteria:

* History of craniofacial surgery or restriction of cervical mobility,
* Edentulous patients
* Pregnancy
* Patients who do not have a proper mouth opening (< 3 cm)
* Patients who might require awake intubation or rapid sequence induction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attending the anesthesiology out-patient clinic for preoperative evaluation in Kanuni Sultan Suleyman Ed. ad Research Hospital. The planned anesthetic method should be general anesthesia.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy | Up to two weeks after preoperative examination
  Grade III or IV laryngeal view before endotracheal intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Avcılar Murat Koluk State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology. 2005 Aug;103(2):429-37. doi: 10.1097/00000542-200508000-00027. PMID 16052126
- [Background] el-Ganzouri AR, McCarthy RJ, Tuman KJ, Tanck EN, Ivankovich AD. Preoperative airway assessment: predictive value of a multivariate risk index. Anesth Analg. 1996 Jun;82(6):1197-204. doi: 10.1097/00000539-199606000-00017. PMID 8638791
- [Background] Apfelbaum JL, Hagberg CA, Caplan RA, Blitt CD, Connis RT, Nickinovich DG, Hagberg CA, Caplan RA, Benumof JL, Berry FA, Blitt CD, Bode RH, Cheney FW, Connis RT, Guidry OF, Nickinovich DG, Ovassapian A; American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2013 Feb;118(2):251-70. doi: 10.1097/ALN.0b013e31827773b2. No abstract available. PMID 23364566
- [Background] Kim JC, Ki Y, Kim J, Ahn SW. Ethnic considerations in the upper lip bite test: the reliability and validity of the upper lip bite test in predicting difficult laryngoscopy in Koreans. BMC Anesthesiol. 2019 Jan 10;19(1):9. doi: 10.1186/s12871-018-0675-5. PMID 30630419
- [Result] Yildirim I, Inal MT, Memis D, Turan FN. Determining the Efficiency of Different Preoperative Difficult Intubation Tests on Patients Undergoing Caesarean Section. Balkan Med J. 2017 Sep 29;34(5):436-443. doi: 10.4274/balkanmedj.2016.0877. Epub 2017 Apr 13. PMID 28443579
- [Result] Selvi O, Kahraman T, Senturk O, Tulgar S, Serifsoy E, Ozer Z. Evaluation of the reliability of preoperative descriptive airway assessment tests in prediction of the Cormack-Lehane score: A prospective randomized clinical study. J Clin Anesth. 2017 Feb;36:21-26. doi: 10.1016/j.jclinane.2016.08.006. Epub 2016 Oct 31. PMID 28183567